CLINICAL TRIAL: NCT05747274
Title: Retrospective Study to Validate the Analytical Performance of an In Vitro Diagnostic (IVD) Medical Device in Patients With Kidney Transplant.
Brief Title: SRDK0921_ Analytical Performance Study
Acronym: SRDK0921_APS
Status: Completed | Type: Observational
Sponsor: BioMAdvanced Diagnostics (Industry)
Collaborators: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SRDK0921_APS
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Kidney Transplant Rejection
Keywords: Gene expression; In Vitro Diagnostic; Subclinical rejection score, kidney allograft

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The Divat COHORT: The DIVAT cohort (Computerized and Validated Data in Transplantation) developed by the Immunology and Nephrology Department of the University Hospital of Nantes (France) , is a biocollection database linked to clinical data and plasma, serum, blood cells and urines of all kidney recipients from Nantes, Paris-Necker, and Lyon centres. The clinical and biological parameters are collected at 3 months, 6 months, 1 year and then every year.
  All available specimens in the DIVAT cohort that:
  * meet inclusion and exclusion criteria of this study AND
  * are usable in terms of quality, integrity, and quantity. will be analysed for this study in order to maximise the power and generalisability of the results.
  Interventions: Device: SRDK0921

INTERVENTIONS:
Device: SRDK0921 — SRDK0921 is an IVD composed of IVD kit for qPCR (SRDK0921KIT) and a cloud-based software (SRDK0921SOFT). It is a class C, rule 3k, IVD according to Regulation (EU) 2017/746.

SUMMARY:
Analytical Performance Study of the SRDK0921 IVD medical device (Kit and Software)

DETAILED DESCRIPTION:
It is a retrospective, observational, non-randomised study using clinical data and samples from DIVAT biocollection.

The aim of this study is to validate the analytical performance of the SRDK0921 In Vitro Diagnostic Medical Device (IVD).

The SRDK0921 system (kit and software) is intended:

* to calculate a score of subclinical rejection in kidney transplant patients
* as an aid in diagnosis of subclinical rejection's absence in kidney transplant recipients in conjunction with other clinical information.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that underwent kidney transplant between January 2008 and January 2016 in the following sites: University hospital center of Nantes, AP-HP Paris-Necker, and HCL Lyon.
* Subjects transplanted from living or deceased donors.
* Patients with an available paired frozen mRNA and biopsy collected at one-year post- transplantation and archived in the DIVAT bio-collection.
* Subjects with good kidney function at one-year post-transplantation (creatininemia below 160 µmol. L-1)
* Subjects under standard immunosuppressive treatments.

Exclusion Criteria:

* Subjects that underwent a graft biopsy for medical indication at one-year post- kidney transplantation.
* Subjects that have stopped immunosuppressive treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples and data from patients included in the DIVAT biocollection are the leftover specimens already used in the Proof-Of-Concept study. All those specimens meet the inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 439 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
AUC (Area Under the Receiver-Operating Characteristic [ROC] Curve) | at 1 year after kidney transplant
  To determine the analytical performance meaning the discriminating ability of the IVD (kit and software), between patients displaying a sub-clinical rejection and patients without subclinical rejection, confirmed with the gold standard method (graft biopsy). An AUC ≥ 0.75 was considered as clinically acceptable.

SECONDARY OUTCOMES:
Analytical sensitivity, specificity, Positive Predictive Value, Negative Predictive Value, Cut-off-value | at 1 year after kidney transplant
  To determine additional indicators of analytical performance of the IVD. PPV: positive predictive value NPV: negative predictive value
Quantification of the gene expression signature | at 1 year after kidney transplant
  To assess the correlation level between the prior Proof-of-Concept study and this study based on the 2 genes expression signature.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Bouler, Study Director — BioMAdvanced Diagnostics
Locations (1):
- Nantes hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided